CLINICAL TRIAL: NCT06705543
Title: Antenatal Investigation of Fetuses With Complex Congenital Heart Defects Using multiOMICS
Acronym: CARDIOMICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/30
Record Dates: First submitted 2024-11-18; First posted 2024-11-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; exome; RNAseq; methylome; biomarkers; environnemental factors; epigenetics
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Congenital Heart Defects population (Active Comparator)
  Interventions: Genetic: multi-omics genetic analyses included exome
- control population (Placebo Comparator)
  Interventions: Genetic: multi-omics genetic analyses

INTERVENTIONS:
Genetic: multi-omics genetic analyses included exome — Genetic analysis will be carried out on amniotic fluid from the volume collected as part of the by obstetricians working in the fetal medicine unit. These genetic analyses will include :
  * Study of free RNA circulating in the LA,
  * Methylome study.
  * Trio exome study (parents-fetus).
  Arms: Congenital Heart Defects population
Genetic: multi-omics genetic analyses — Genetic analysis will be carried out on amniotic fluid from the volume collected as part of the by obstetricians working in the fetal medicine unit; These genetic analyses will include :
  * Study of free RNA circulating in the LA,
  * Methylome study.
  Arms: control population

SUMMARY:
This study will use multiOMICS study on fetuses with complexe congenital heart defects (CHD) to identify etiological epigenetic factors of these cardiac malformations, related to environmental factors during pregnancy.

DETAILED DESCRIPTION:
Congenital heart defects (CHDs) are a very heterogeneous group of heart diseases in terms of embryonic mechanisms, phenotypes and aetiologies. In isolated forms, genetic causes are identified in only 19% of cases, linked to chromosomal abnormalities (8%) or gene variants (11%). Environmental causes such as infection, exposure to toxic substances or ingestion of teratogenic substances may also favour the onset of MCC. Although in the majority of cases the aetiology remains unknown, the discovery of MCC in the ante-natal period almost systematically leads to a genetic aetiological work-up using amniotic fluid for karyotype, Array-CGH and, more recently, exome analysis. With regard to environmental causes, recent data in the literature report a link between environmental exposures (occupational, extra-occupational or medicinal) and congenital anomalies.

Objectives: The low percentage of genetic abnormalities and toxic factors identified as causal in patients with non-syndromic CHD prompts a search for more complex causes such as epigenetic modifications linked to an interaction between genes and environmental factors.

Methods: The multi-omics study approach, using high-throughput sequencing technologies (exome, RNASeq, methylSeq), provides a wealth of information on cellular and/or tissue signaling pathways in response to exposure. Integrated analysis of transcriptomes and methylomes has demonstrated the occurrence of combined defects in gene expression and methylation following toxic exposure. The period of CHD formation during embryonic development prompts us to look for epigenetic modifications during prenatal period, as close as possible to the pathophysiological mechanisms leading to this malformation.

Expected results: the multi-omics analysis applied to fetuses with non-syndromic complex CHD, combined with the characterization of occupational and non-occupational environmental exposures, will enable us to extend the etiological search for these malformations, to identify biomarkers linked to the occurrence and severity of these malformations and gain a better understanding of the pathophysiological mechanisms linked to CHD.

In the longer term, this study will serve as a basis for large-scale studies to enable the development of prevention policies, based on exhaustive, multicenter cohorts. In addition, multi-omics studies could identify gene markers, by exome, transcriptome and/or methylome, which could then be studied in a targeted manner.

ELIGIBILITY:
Inclusion Criteria:

Fetuses with congenital heart disease :

* Pregnant women aged 18 and more
* Single foetal pregnancy in which the foetus has a complex non-syndromic congenital heart defect, with no identified chromosomal abnormality, gene syndrome or infection.
* Patient for whom the indication for amniocentesis has been accepted by the CPDPN and accepted by the couple/patient
* Gestational age between 20 and 28 weeks' gestation.
* Person affiliated to or benefiting from a social security scheme.
* Free, informed and express consent (confirmed in writing) (at the latest on the day of inclusion and before any examination required by the research).

Control Population for RNAseq and MéthlySeq

* Pregnant women aged 18 and more
* Patient in whom the indication for amniocentesis has been retained by the CPDPN and accepted by the couple/patient, for a non-malformative ultrasound anomaly (hyperechoic bowel, idiopathic hydramnios, increased risk of trisomy 21, agenesis of the OPN, suspected toxoplasmosis/CMV seroconversion), with no chromosomal anomaly, gene syndrome or infection identified.
* Gestational age between 20 and 28 weeks' gestation.
* Person affiliated to or benefiting from a social security scheme.
* Free, informed and express consent (confirmed in writing) (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

For both populations (cases and controls) :

* Female minors,
* Patients not affiliated to the social security system,
* Patients who do not understand French,
* Patients under guardianship
* Multiple pregnancies, or where the foetus has associated malformations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac malformations biomarkers | Visit 1 : day 0
  Identification of biomarkers such as RNA deregulation (mRNA, LncRNA, miRNA, upregulated or deregulated compared to controls), and DNA methylation marks (present or absent, compared to controls) specific to cardiac malformations by transcriptomic and methylomic analysis of amniotic fluid from fetuses with congenital heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROORYCK-THAMBO, PROF, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No